CLINICAL TRIAL: NCT02298283
Title: Brentuximab Vedotin as Consolidation Treatment in Patients With Stage I/II Hodgkin's Lymphoma and FDG-PET Positivity After 2 Cycles of ABVD
Brief Title: Brentuximab Vedotin as Consolidation Treatment in Patients With Stage I/II HL and PET Positivity After 2 Cycles of ABVD
Acronym: BRAPP2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRAPP2
Record Dates: First submitted 2014-11-13; First posted 2014-11-21 (Estimated); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin lymphoma; HL; brentuximab vedotin
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Cyclophosphamide; Doxorubicin; Vincristine; Bleomycin; Etoposide; Procarbazine; Prednisone; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- study treatment (Experimental): * induction = BEACOPP-escalated (bleomycin, etoposide, adriamycin, cyclophosphamide, oncovin, procarbazine, and prednisone) : 2 cycles every 3 weeks
  * radiotherapy = involved field radiotherapy (IFRT) will be given 3 to 4 weeks after the last day of second BEACOPP at 30 Grays (+boost 6 Grays to area with residual lesion) in 3 weeks
  * Consolidation = brentuximab vedotin treatment will start 4 weeks after the last day of IFRT and up to 6 weeks. The dose of study treatment is 1.8 mg/kg
  Interventions: Drug: brentuximab vedotin; Drug: Cyclophosphamide; Drug: Adriamycin; Drug: Oncovin; Drug: Bleomycin; Drug: Etoposide; Drug: Procarbazine; Drug: Prednisone; Drug: G-CSF; Radiation: 30 Grays

INTERVENTIONS:
Drug: brentuximab vedotin — is 1.8 mg/kg administrated by IV infusion
  Other Names: SGN35
Drug: Cyclophosphamide — 1250 mg/m², IV, part of the BEACOPP chemiotherapy, D1 of 2 BEACOPP cycles, every 3 weeks
Drug: Adriamycin — 35mg/m², IV, part of the BEACOPP chemiotherapy, D1 of 2 BEACOPP cycles, every 3 weeks
  Other Names: Doxorubicin
Drug: Oncovin — 1.4 mg/m², IV, part of the BEACOPP chemiotherapy, D8 of 2 BEACOPP cycles, every 3 weeks
  Other Names: Vincristin
Drug: Bleomycin — 10 mg/m², IV, part of the BEACOPP chemiotherapy, D8 of 2 BEACOPP cycles, every 3 weeks
Drug: Etoposide — 200 mg/m², IV, part of the BEACOPP chemiotherapy, D1 to D3 of 2 BEACOPP cycles, every 3 weeks
Drug: Procarbazine — 100 mg/m², IV, part of the BEACOPP chemiotherapy, D1 to D7 of 2 BEACOPP cycles, every 3 weeks
Drug: Prednisone — 40 mg/m², IV, part of the BEACOPP chemiotherapy, D1 to D7 of 2 BEACOPP cycles, every 3 weeks
Drug: G-CSF — 5 µg/kg/j, SC, D9 until GB 1.0x109/L
Radiation: 30 Grays — 30 Gy radiation of sites initially diagnoses + 6Gy for residual sites, 3 to 4 weeks after D1 of BEACOPP cycle 2.

SUMMARY:
This study aims to evaluate the efficacy brentuximab vedotin as consolidation treatment in patients with stage I/II Hodgkin's lymphoma and 18-fluorodeoxyglucose (FDG) -PET positivity after 2 cycles of ABVD (adriamycin, bleomycin, vinblastine, and dacarbazine).

DETAILED DESCRIPTION:
This study aims to evaluate the progression free survival after treatment for patient with stage I/II supradiaphragmatic HL patient and PET positive after 2 courses of ABVD.

The treatment consist of 3 phases :

* induction treatment with 2 cycles every 3 weeks of bleomycin, etoposide, Adriamycin, cyclophosphamide, oncovin, procarbazine, and prednisone (BEACOPP) escalated
* radiotherapy 30 Gy starting 3 to 4 weeks after last day of second course of BEACOPP-escalated
* consolidation treatment with 8 cycles every 21 days of brentuximab vedotin

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed cluster of differentiation antigen 30+ (CD30+) classical Hodgkin lymphoma
2. Patients must have provided voluntary written informed consent
3. Supradiaphragmatic Ann Arbor clinical stage I or II
4. Mandatory PET scan performed at diagnosis
5. Patients treated with first-line ABVD and PET scan positive after 2 cycles (Deauville score 4 & 5)
6. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
7. Life expectancy > 6 months
8. Patients must be 18-65 years of age
9. Patients must be available for periodic blood sampling, study-related assessments and management of toxicity at the treating institution
10. Female patients who:

    * Are postmenopausal for at least 1 year before the screening visit OR are surgically sterile OR
    * If they are of childbearing potential, agree to practice 2 effective methods of contraception at the same time
11. Male patients, even if surgically sterilized, who agree to practice effective barrier contraception during the entire study treatment period and through 6 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse
12. Clinical laboratory values as specified below before the first dose of study drug:

    * Absolute neutrophil count ≥ 1,500/µL
    * Platelet count ≥ 75,000/ µL
    * Total bilirubin must be < 1.5 x the upper limit of the normal (ULN) unless the elevation is known to be due to Gilbert syndrome
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST)must be < 3 x the upper limit of the normal range
    * Serum creatinine must be < 2.0 mg/dL and/or creatinine clearance or calculated creatinine clearance > 40 mL/minute
    * Hemoglobin must be ≥ 8g/dL
13. Patient affiliated to social security system

Exclusion Criteria:

1. Patients with dementia or altered mental status that would preclude compliance with drug delivery
2. Women who are pregnant or breastfeeding
3. Patients with symptomatic pulmonary disease
4. Patients with known history of any of the following cardiovascular conditions:

   * Myocardial infarction within 2 years of inclusion
   * New York Heart Association (NYHA) Class III or IV heart failure
   * Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
   * Recent evidence (within 6 months before first dose of study drug) of a left-ventricular ejection fraction <50%
5. Any history of cancer or cancer treatment during the last 3 years with the exception of non-melanoma skin cancer or stage 0 (in situ) carcinoma of any type if they have undergone complete resection
6. Uncontrolled infectious disease, including active Hepatitis B Virus (HBV) infection defined by either detection of Hepatitis B surface (HBs) Antigen or presence of Hepatitis B core (HBc) antibody without detectable anti HBs antibody
7. Any active systemic viral, bacterial, or fungal infection requiring systemic antibiotics at the time of inclusion and planned to be still on going within 2 weeks prior to first study drug dose
8. Known Human Immunodeficiency Virus (HIV), known or suspected hepatitis C Virus (HCV) or human T-cell lymphotrophic virus (HTLV) serology positivity
9. Patients who have been treated previously with any anti-CD30 antibody
10. Known hypersensitivity to any excipients contained in the brentuximab vedotin formulation
11. Known cerebral or meningeal disease (HL or any other etiology), including signs or symptoms of Progressive Multifocal Leukoencephalopathy (PML)
12. Any sensory or motor peripheral neuropathy greater than or equal to Grade 2
13. Patients that have not completed any prior treatment chemotherapy and/or other investigational agents within at least 5 half-lives of last dose of that prior treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2 years
  PFS is defined as the time from the date of the first cycle of ABVD to the first observation of documented disease progression or death due to any cause.

SECONDARY OUTCOMES:
Complete Response rate (CR rate) | 35 weeks
  according to Cheson 2007
Overall survival | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Pauline BRICE, MD, Principal Investigator — Lymphoma Study Association; Thomas GASTINNE, MD, Principal Investigator — Lymphoma Study Association
Locations (30):
- France (30):
  - CH Victor Dupouy, Argenteuil
  - Polyclinique Bordeaux Nord, Bordeaux
  - Centre François Baclesse, Caen
  - CH de Chambéry, Chambéry
  - CH Sud Francilien, Corbeil-Essonnes
  - Hôpital Henri Mondor, Créteil
  - CHU de Dijon - Hôpital le Bocage, Dijon
  - Hôpital André Mignot, Le Chesnay
  - Clinique Victor Hugo, Le Mans
  - CHRU Lille - Hôpital Claude Huriez, Lille
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmette, Marseille
  - Hôpital de la Conception, Marseille
  - CHU Montpellier - Saint ELOI, Montpellier
  - CHU de Nantes, Nantes
  - Hôpital Cochin, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital de la Pitié Salpétrière, Paris
  - CH Perpignan, Perpignan
  - Hôpital Haut Lévêque, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - CHU Robert Debre, Reims
  - CHU Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - CHU de Strasbourg, Strasbourg
  - I.U.C.T Oncopole, Toulouse
  - CHU Bretonneau, Tours
  - CHU de Brabois, Vandœuvre-lès-Nancy
  - Gustave Roussy Cancer Campus, Villejuif

IPD SHARING:
Plan to Share IPD: No